CLINICAL TRIAL: NCT05600608
Title: Augmentation of Volatile Biomarkers of Oesophageal and Gastric Adenocarcinoma From the Tumour Lipidome
Acronym: AVOCADO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anuja Mitra (Other)
Collaborators: British Medical Research Council (Other Government); British Association of Surgical Oncology (Unknown); The Royal College of Surgeons of England (Other)
Responsible Party: Sponsor-Investigator, Anuja Mitra, Dr, MRC Clinical Research fellow, Imperial College London
Organization: Imperial College London (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21HH6980
Record Dates: First submitted 2022-10-25; First posted 2022-10-31 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Breath Test; Oesophageal Cancer; Gastric Cancer; Augmentation; Diagnoses Disease
Keywords: volatile organic compounds; breath test; augmentation; lipid; oesophageal cancer; gastric cancer; non- invasive
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: All study participants will receive the same formulation, dose and amount of the oral stimulant drink. Breath samples will be taken at baseline and then at the same time points following consumption of the drink.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oesophago- gastric adenocarcinoma patients (Experimental): Oesophagogastric adenocarcinoma (OG) cancer patients (who are neoadjuvant chemotherapy treatment naïve) will receive 120mls of a sterile oral stimulant drink (OSD) (manufactured by Ingenza ltd), which is an ISO accredited laboratory. The active component of the drink is iron sulphate (5g/l), pH 5-6.
  Breath will be taken following an optimised methodology designed by the VOC laboratory at Imperial college London at baseline and then at 30, 60 and 90 minutes following consumption of the drink.
  Participants will be nil by mouth for 6 hours prior to the breath test, they can have water up to 2 hours before the breath test.
  Interventions: Dietary Supplement: Oral Stimulant Drink
- Benign healthy control patients (Active Comparator): Age, gender and demographic matched patients who have had a negative oesophagogastroscopy within 1 year which is negative for adenocarcinoma will be recuited into the comparison arm. Patients will be given the same OSD and breath will be sampled at the same time points as the experimental arm.
  Interventions: Dietary Supplement: Oral Stimulant Drink

INTERVENTIONS:
Dietary Supplement: Oral Stimulant Drink — please see description of the drink in the arm/ group section

SUMMARY:
Nearly 10,000 people die each year in the United Kingdom from cancer of the lower gullet and stomach, known as known as oesophago- gastric adenocarcinoma (OGC). OGC is detected late as symptoms are non- specific and often mistaken for common problems such as heartburn. This translates to fewer than 2 in every 10 patients diagnosed with OGC living longer than 5 years.

The breath of people with OGC is enriched with volatile chemicals (VOCs) that indicate cancer. When measured in a breath test, it detects OAC 80 out of 100 times. Whilst encouraging, there is scope to improve the detection rate by giving patients a stimulant drink that amplifies the production of tumour specific VOCs only, to increase their detection in the breath test.

The goal of this observational study is to produce an enhanced second-generation breath test with superior ability to detect OGC through augmentation of breath. This will improve long term survival from cancer using an entirely non- invasive test.

All participants (cancer and control participants) will consume an oral stimulant drink (OSD) and provide breath samples pre and post consumption of the drink at set time points (maximum 2 hours after consumption of the drink).

The investigators will compare the breath VOCs from both groups, before and after consumption of the OSD to see if the OSD has a desired augmentation effect and can improve the accuracy of the OGC breath test.

With this second-generation breath test, participants with vague symptoms can undergo a quick, non- invasive test, have samples analysed in a safe and accurate manner and be subsequently stratified based on their risk of having OGC, leading to earlier disease detection and improved clinical outcomes.

DETAILED DESCRIPTION:
Introduction: Early detection of oesophago- gastric adenocarcinoma (OGC) with improved diagnostics is essential to reduce the burden of this aggressive cancer. The breath of people with OAC is enriched with volatile organic compounds (VOC). A breath test based on these VOCs has an 80% sensitivity and 81% specificity of detecting OAC. The diagnostic accuracy may be further improved by using an exogenous stimulant that amplifies the production of OGC specific VOCs. This strategy is known as 'augmentation'. It is possible to compare intra- subject breath (pre and post stimulant) and use the fold increase in VOCs to detect cancer. This is the investigator's novel approach to improving breath test sensitivity and early OGC detection. The biology of the OGC VOCs must be first understood to selectively augment their production.

Background: The OGC lipidome is enriched with phospholipids that are vulnerable to degradation via lipid peroxidation, which is a principal mechanism for endogenous VOC production. Prokaryotic lipids in the OGC microbiome are also vulnerable to peroxidation. Putative drivers of lipid peroxidation are higher in tumour environment. This suggests OGC lipids and/ or prokaryotic lipids may be source compounds for diagnostic VOCs and this mechanism may be augmented.

Aim: to augment the production of OGC VOCs to improve the diagnostic performance of the breath test.

Proposal: 1) A lipidomics study of the onco- microbial lipidome using bespoke mass spectrometry with phenotyping of the corresponding VOCs will identify source lipids that generate diagnostic VOCs, 2) data driven stable isotope experiments to select an augmentation model based on the degradation kinetics of the source lipid in vivo and 3) translating the science to clinic with a study of the augmented breath test in participants with OGC.

Translation of the novel scientific data generated to clinic presents a real opportunity to improve clinical outcomes in people with OGC.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be over 18 years old and up to the maximal age of 90 years , AND:
* Have a confirmed histological diagnosis of oesophageal OR gastric adenocarcinoma at Imperial NHS Healthcare Trust, AND
* Will undergo am oesophagogastroscopy (OGD) as part of their routine clinical care, OR:
* Will undergo surgical resection of their oesophageal or gastric cancer as part of their routine clinical care OR
* Any patient with non- cancerous upper gastrointestinal (benign) problem who will have an OGD OR surgery as part of their routine clinical care at Imperial NHS Trust

Exclusion Criteria:

* Participant that lacks capacity or is unable to provide informed consent
* Any participant below 18 years of age or over 90 years of age
* Participants with allergies to any aspect of the metabolic drink
* Participants who have had previous OG surgical resection

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
To establish a second- generation augmented breath test with improved diagnostic accuracy for the detection of OG adenocarcinoma. | 12 months
  This breath test will utilise serial breath sampling following the ingestion of an augmentation solution (OSD). Breath samples will be taken pre and post consumption of the OSD and fold changes in the VOCs will be calculated. The entire process of breath sampling is non- invasive.
To determine the diagnostic accuracy of the augmented exhaled breath test, in the prediction of oesophago-gastric cancer (OGC). | 12 months
  The investigators will generate an untargeted VOC breath model following exhaled VOC augmentation.

SECONDARY OUTCOMES:
To comprehensively characterise the tissue lipid input and lipidomic reprogramming in oesophagaeal and gastric adenocarcinoma in comparison to healthy non- cancer tissues. | deadline December 2022
  Liquid chromatography mass spectrometry (LCMS) comprehensive lipidomic OGC tissue profiling will be performed by the investigators to generate a lipid map in healthy and cancer tissues.
To identify the mechanistic pathways and origins of the production of breath Volatile compounds by investigating the tumour lipidome. | 12 months
  The investigators will perform a range of in silico, in vitro and ex vivo experiments that determine the mechanisms and kinetics of lipid to VOC generation

CONTACTS AND LOCATIONS:
Overall Officials: George B Hanna, FMedSci, Principal Investigator — Imperial College London
Locations (1):
- Volatile Biomarker Group, Commonwealth Building, Hammersmith Hospital, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Metabolomic and experimental data will be shared as participants will be given a unique identifier rendering the information anonymous. All other data collated will be stored in a central secure repository under an embargo and will be suitable for sharing following approval by the Chief Investigator.
  New users can access a simple study policy and summarised data on the Imperial Clinical Research Network study website. Research data will also be discovered on the NIHR In-Vitro Diagnostic Co-operative website. Data will be disseminated through presentation at leading conferences that are accessible to subject specific and generalist audiences. Publication in high impact journals will allow global discovery of data to new users.
  Decisions to supply research data to new users will be made by: Dr Anuja Mitra, Professor Griffin and Professor Hanna (PI).
Supporting Information: Study Protocol, CSR
Time Frame: 3 years after the study has completed recruitment (December 2026). The information will be available for sharing for 2 years after that (until December 2028).
Access Criteria: Decisions to supply research data to new users will be made by: Dr Anuja Mitra, Professor Griffin and Professor Hanna (PI).
URL: http://london.ivd.nihr.ac.uk/

REFERENCES:
- [Background] Mitra A, Choi S, Boshier PR, Razumovskaya-Hough A, Belluomo I, Spanel P, Hanna GB. The Human Skin Volatolome: A Systematic Review of Untargeted Mass Spectrometry Analysis. Metabolites. 2022 Sep 1;12(9):824. doi: 10.3390/metabo12090824. PMID 36144228
- [Result] Markar SR, Wiggins T, Antonowicz S, Chin ST, Romano A, Nikolic K, Evans B, Cunningham D, Mughal M, Lagergren J, Hanna GB. Assessment of a Noninvasive Exhaled Breath Test for the Diagnosis of Oesophagogastric Cancer. JAMA Oncol. 2018 Jul 1;4(7):970-976. doi: 10.1001/jamaoncol.2018.0991. PMID 29799976
- [Result] Antonowicz S, Bodai Z, Wiggins T, Markar SR, Boshier PR, Goh YM, Adam ME, Lu H, Kudo H, Rosini F, Goldin R, Moralli D, Green CM, Peters CJ, Habib N, Gabra H, Fitzgerald RC, Takats Z, Hanna GB. Endogenous aldehyde accumulation generates genotoxicity and exhaled biomarkers in esophageal adenocarcinoma. Nat Commun. 2021 Mar 5;12(1):1454. doi: 10.1038/s41467-021-21800-5. PMID 33674602